CLINICAL TRIAL: NCT03567395
Title: Honey to Improve Sleep Quality: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jane Alcorn, Associate Dean Research and Graduate Affairs, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIO 018-31
Record Dates: First submitted 2018-04-22; First posted 2018-06-25 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Poor Quality Sleep
MeSH Terms: interventions — Melatonin; Honey

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator): Melatonin (5 mg sublingual tablet)
  Interventions: Dietary Supplement: Melatonin
- Honey (Experimental): raw honey (1.5 tablespoons)
  Interventions: Dietary Supplement: Honey

INTERVENTIONS:
Dietary Supplement: Melatonin — Melatonin (5 mg sublingual tablet) administered for 3 days
  Arms: Melatonin
Dietary Supplement: Honey — Raw Honey (1.5 tablespoons) administered for 3 days
  Arms: Honey

SUMMARY:
Inadequate sleep quality and duration may result in adverse health outcomes and poorer quality of life. Despite the availability of behavior modification and pharmaceuticals to aid sleep optimization and quality approximately 50% men and women continue to experience difficulty falling asleep or staying asleep. Individuals with sleep disorders may find adherence to such interventions difficult to maintain (e.g. behavior modification) or the therapies may pose a risk (e.g. dependence on pharmaceuticals). A need exists for alternative therapeutic interventions, particularly those that are simple and cost effective. Observational and anecdotal data supports honey as a functional food to promote better sleep. As an initial step towards developing an evidence base for honey for improvement of sleep quality the investigators propose to conduct a preliminary open-label proof-of-principle study to assess the feasibility (primary outcome) and potential effectiveness (secondary outcome) of honey in improving sleep quality before embarking upon a full-scale pivotal clinical trial. The study data will confirm safety of honey use in a population of poor sleepers and to identify where improvements in study design are necessary in planning of a larger clinical trial.

DETAILED DESCRIPTION:
The feasibility study will involve an open-label, crossover study with 20 participants (Age 18 - 55; 10 male, 10 female) in a population-based setting meeting the inclusion criteria and giving informed consent. As a feasibility study, the investigators did not conduct a power analysis and sample size is typical of other feasibility studies. To control for possible differences in sex, an equal number of male and female participants will be recruited. Participants will be recruited from clients of the Medicine Shoppe Pharmacy (Place Riel) and invited to participate through their interaction with the study pharmacists (Carla Guedo or Amber Ly) or by poster advertisement posted at the participating pharmacy or posted around the university and on PAWS. Prospective participants will undergo a screening to determine suitability for inclusion into the trial using an adaptation of the PharmaZZZ screening form (see attached document). Prior to the initiation of the treatment arms, consented participants will have baseline characteristics collected (sex, age, body weight, smoking status, socio-professional status). Furthermore, consented participants will complete a screening form (modified from the PharmaZZZ program, see attachment) and an Insomnia Severity Index (see attachment).

For the intervention, participants will be instructed to limit consumption of coffee, black tea, alcohol, energy drinks, and other caffeinated products one week before and during the treatment and washout periods. The interventions are raw honey (1.5 tablespoons) or melatonin (5 mg sublingual tablet). To randomize sequence of treatment and participants, the investigators will employ a randomization table in a standard statistical textbook. Three days prior to the treatment intervention, participants will be asked to eat supper at approximately 6 pm and maintain a consistent intake of macronutrients for each supper meal. A nutritionist will be consulted to help plan supper meals. During this 3 day period participants will complete a daily sleep hygiene Log (see attachment) and morning sleep log (see attachment), which assesses subjective measures of sleep quality and amount. On the fourth day participants will continue the daily sleep hygiene log and sleep log, and evening meal pattern, but will take either melatonin or honey by mouth within 30 minutes of going to sleep for three consecutive days. At the end of the 3 day treatment period, participants will discontinue with the sleep logs and prescriptive meal pattern and resume usual activities during a 7 day washout between treatment arms. Participants also will be asked to complete a Leeds Sleep Evaluation Questionnaire (LSEQ) (see attachment, slightly modified from published questionnaire), a standardized self-reporting instrument that assesses ease of getting to sleep (questions 1 - 3), the quality of sleep (questions 4, 5), awakening from sleep (questions 6, 7), and behavior following wakefulness (questions 8 - 10) in the morning of day 4 and day 7 of the treatment arm. LSEQ is considered a sensitive indicator of how the subject perceives or feels changes in sleep quality and latency. At the end of the washout, participants will repeat the cycle with the alternative treatment (i.e. 3 days prior to the treatment intervention, participants will be asked to eat supper at 6 pm, maintain a consistent intake of macronutrients for each supper meal, complete a daily sleep hygiene log and sleep log, begin alternative treatment on fourth day for 3 days, and then discontinue with the sleep logs and prescriptive meal pattern, complete LSEQs, and resume usual activities). The investigators will provide participants with a visual schedule (calendar) to follow to ensure that each understands the requirements of the study.

The honey will be Canada #2 White Honey from SweetHeart Pollinators (Janeil Enterprises, Eatonia, SK). Melatonin (5 mg sublingual tablet; McKesson) will be dispensed by the participating pharmacists (Carla Guedo or Amber Ly). Each treatment requires that the dispensing pharmacist place an appropriate volume of the treatments into individual disposable condiment containers with lids using aseptic techniques. An individual appropriately labeled container for each treatment day will be made available to the participants. The treatments will be known to the participant and study personnel. All used and unused containers will be returned to the pharmacist to assess compliance. The pharmacist will maintain accurate records of all treatments dispensed with identification of the participant to whom they were dispensed, date of dispensing, and unused treatments. Each participant will obtain the study's supply of each treatment (3 containers/treatment) in larger plastic bags labelled as "Study Treatment honey or melatonin" with dosing instructions (e.g. using a teaspoon consume the entire contents of the container once daily within 30 minutes of going to sleep and follow with a small glass of water). The participant will return to the pharmacy all used and unused containers as well as completed logs and questionnaires to the pharmacy at the end of the study period.

For evaluation of sleep quality, criteria will be the monitoring of participant perception of sleep quality by using the morning sleep logs and the LSEQ. Stopping rules or discontinuation criteria for a participant includes violation of exclusion criteria and non-compliance with the protocol. Participants will also be free to voluntarily withdraw from the study at any time. If a participant withdraws, no further data will be collected from the participant. The subjective variables of sleep quality will be assessed using repeated measures analysis of variance (ANOVA). Other variables of interest will be analyzed using a student's t-test for continuous variables and Fisher's exact test for categorical variables. Patient demographic data and subjective sleep variables will be reported descriptively as means and standard deviations.

ELIGIBILITY:
Inclusion Criteria:

Age: 18 - 55

* Male or female
* Able to comply with study protocol and give informed consent
* Healthy (no diagnosis of medical or mental illness) (not suffering from vascular disease, diabetes mellitus, hyperlipidemia, obesity (body mass index over 30), dermatological disease, gynecological disease, endocrine disease)
* Discontinuation of sleep aids 4 weeks in advance of the study
* Self-report of having difficulty sleeping for 1 week or more

Exclusion Criteria:

* Age: <18 and >55

  * Type I and Type II diabetes, current infectious disease (e.g. cold or flu)
  * Unstable medical condition
  * History of psychiatric disorder (past or present)
  * Pain syndrome affecting sleep
  * Obese (BMI over 30)
  * Pregnant or lactating women
  * Lifestyle habits that would modify the wake-sleep rhythm (e.g. night work; shift work; young children that interrupt sleep)
  * Substance and/or drug dependence (alcohol, nicotine, pain killers)?
  * Use of the following medications during the study period: oral or injectable corticosteroid, sedating antihistamines (e.g. cold, allergy, motion sickness), psychotropic medications or hypnotics, benzodiazepine, narcotics, any illicit drugs
  * Use of stimulants (>4 cups (1 cup = 250 mL) of coffee/day)
  * Participation in any other clinical trial with an investigational agent within one month prior to randomization

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Completion of sleep hygiene log | 2 weeks
  Feasibility of participants to be compliant to a required sleep quality measurement tool, the sleep hygiene log
Completion of morning sleep log | 2 weeks
  Feasibility of participants to be compliant to a required sleep quality measurement tool, the morning sleep log
Completion of Leeds Sleep Evaluation Questionnaire | 2 weeks
  Feasibility of participants to be compliant to standardized assessment tool of sleep quality, the Leeds Sleep Evaluation Questionnaire. This questionnaire consists of 10 questions with a scale from 1 - 9, the highest number for each symptom measured representing the best sleep quality. Score of 5 is the baseline such that a score of 5 indicates no change and a higher or lower value from 5 indicates a change in a symptom. A total score will be reported to determine whether the intervention resulted in a change in sleep quality.

SECONDARY OUTCOMES:
Sleep quality as measured by daily sleep hygiene log | 6 days
  Assessment of the quality of sleep as measured by a daily sleep hygiene log, which assesses subjective measures of sleep quality and amount by the end of the 3 day intervention with the treatments (honey or melatonin)
Sleep quality as measured by daily morning sleep log | 6 days
  Assessment of the quality of sleep as measured by a daily morning sleep log, which assesses subjective measures of sleep quality and amount by the end of the 3 day intervention with the treatments (honey or melatonin)
Sleep quality as measured by Leeds Sleep Evaluation | 6 days
  Assessment of the quality of sleep as measured by a standardized tool, the Leeds Sleep Evaluation Questionnaire), which assesses subjective measures of sleep quality and amount, by the end of the 3 day intervention with the treatments (honey or melatonin)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Alcorn, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- Medicine Shoppe, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No